CLINICAL TRIAL: NCT06267014
Title: Use of a Virtual Reality Cognitive Stimulation Programme for Breast Cancer Patients Wishing to Restart or Maintain a Professional Activity
Acronym: Cog-RV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-A02163-42
Record Dates: First submitted 2024-02-09; First posted 2024-02-20 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer; Cancer-related Cognitive Difficulties
Keywords: virtual reality; cognitive rehabilitation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients will follow the Virtual Reality program developed for the study, during the cognitive rehabilitation sessions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Reality sessions (Experimental)
  Interventions: Behavioral: Virtual Reality sessions

INTERVENTIONS:
Behavioral: Virtual Reality sessions — One session during 10-15 minutes per week for 6 weeks.

SUMMARY:
The study concerns patients who have been treated for breast cancer, have cognitive problems and are planning to return to work or are currently working and wish to begin cognitive rehabilitation.

Patients will follow the Virtual Reality program developed for the study, during the cognitive rehabilitation usually proposed in the establishment, at the rate of a weekly session of 10-15 minute for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years of age
* Patient with breast cancer for whom adjuvant chemotherapy has been administered; maintenance treatments (e.g. Trastuzumab, hormone therapy) are eligible,
* Maximum 2 years after completion of adjuvant treatment,
* Patients who have cognitive complaints at inclusion (answer yes to the question: 'Since your cancer treatment, have you had any difficulties with memory, concentration, etc.?)
* Patients planning to return to work or who have returned to work in the past year,
* Signature of informed consent prior to any specific procedure relating to the study,
* Patient affiliated to a social security system.

Exclusion Criteria:

* Patients suffering from illnesses or conditions that impair their ability to understand, follow and/or comply with study procedures,
* Patients with personality disorders and/or psychiatric pathology,
* Patients deprived of their liberty or placed under the authority of a guardian,
* Pregnant women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2024-05-23 (Actual); Primary Completion 2026-02-06 (Actual); Study Completion 2026-02-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients adhering to the Virtual Reality program | At 6 weeks
  Adherence is defined as the completion of at least 5 of the 6 sessions planned.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre François Baclesse, Caen, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vieira Jales I, Hummel E, Clarisse B, Gouranton V, Cogne M, Lecuyer A, Leconte A, Lequesne J, Ahmed-Lecheheb D, Morel A, Fernette M, Joly F, Lange M. Virtual reality-based cognitive rehabilitation programme to support employment in patients with breast cancer: protocol for the Cog-RV pilot study. BMJ Open. 2025 Dec 15;15(12):e112196. doi: 10.1136/bmjopen-2025-112196. PMID 41401994